CLINICAL TRIAL: NCT04039035
Title: Preoperative Nutritional Assessment of The Patients Undergoing Major Gastrointestinal Surgery and Their Immediate Postoperative Outcome
Status: Completed | Type: Observational
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Nabin Pokharel, Assistant Professor/ Senior Medical Officer, National Academy of Medical Sciences, Nepal
Other Study IDs: 788/2072/73
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Preoperative Nutritional Status and the Postoperative Outcome
Keywords: Nutritional Risk Index; Body mass Index; Postoperative Complications; Length of Hospital Stay and Cost.
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It was a prospective observational study, where preoperative nutritional status and early postoperative complications <30 days (infectious or noninfectious) were studied. The patients admitted between July 2015 to May 2017, who underwent major GI surgeries were included in the study. The study was designed to check if BMI and NRI can predict the postoperative outcomes in these patients.

DETAILED DESCRIPTION:
It was a prospective observational study. This study was done at NAMS, Bir Hospital, Kathmandu, Nepal between July 2015 to May 2017. All the patients who underwent major GI surgery, under general anesthesia, were included in the study. Major was defined as surgery involving >2hrs and excluded were an emergency major operation, gallstone disease operations, patients with cough, fever, and chest infections respectively. The sample size was calculated using the formula z2pq/d2. Twice the number of sample calculated was taken into consideration and the maximum tolerable error was taken as 5%. BMI and NRI were two independent categorical variables. The dependent variables were the postoperative outcome in terms of infectious and noninfectious complications. All the preoperative parameters were of the patients were recorded. The immediate postoperative complications were documented and categorized as infectious and noninfectious complications.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who underwent major GI surgery, under general anesthesia, were included in the study. Major was defined as surgery involving >2hrs and

Exclusion Criteria:

* Excluded were an emergency major operation, gallstone disease operations, patients with cough, fever, and chest infections respectively

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patient who underwent major GI surgery in NAMS Bir Hospital (a tertiary level hospital of Government of Nepal) between 2015 to 2017.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Infectious and noninfectious complication | 3 years
  Correlation between NRI/BMI and postoperative complications (infectious and noninfectious). The NRI is calculated using the formula: NRI = (15.9 × serum albumin g/L) + (41.7 × current weight/usual weight). The usual weight was defined as the stable weight 6 months before the illness in Kilograms. NRI > 100 indicated that the patient is not malnourished, while 97.5-100 indicated mild malnourishment, 83.5-97.5 indicated moderate malnourishment and <83.5 indicated severe malnourishment respectively. And BMI is defined as the weight in Kilograms divided by the square of height in Meters.

SECONDARY OUTCOMES:
Length of hospital stay and cost | 3 years
  NRI and BMI may predict the length of hospital stay and cost

CONTACTS AND LOCATIONS:
Overall Officials: Nabin Pokharel, MCh, Principal Investigator — NAMS, Bir Hospital
Locations (1):
- Department of Surgical Gastroenterology, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
We may share the datas if there is an interest from other researcher group. At present it is undecided.

REFERENCES:
- [Result] Soeters P, Bozzetti F, Cynober L, Forbes A, Shenkin A, Sobotka L. Defining malnutrition: A plea to rethink. Clin Nutr. 2017 Jun;36(3):896-901. doi: 10.1016/j.clnu.2016.09.032. Epub 2016 Oct 8. PMID 27769782
- [Result] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Result] Pereira TG, da Silva Fink J, Silva FM. Thickness of the adductor pollicis muscle: Accuracy in predicting malnutrition and length of intensive care unit stay in critically ill surgical patients: Thickness of the adductor pollicis muscle in surgical critically patients. Clin Nutr ESPEN. 2018 Apr;24:165-169. doi: 10.1016/j.clnesp.2017.10.013. Epub 2018 Feb 15. PMID 29576356
- [Result] Jensen GL, Mirtallo J, Compher C, Dhaliwal R, Forbes A, Grijalba RF, Hardy G, Kondrup J, Labadarios D, Nyulasi I, Castillo Pineda JC, Waitzberg D; International Consensus Guideline Committee. Adult starvation and disease-related malnutrition: a proposal for etiology-based diagnosis in the clinical practice setting from the International Consensus Guideline Committee. JPEN J Parenter Enteral Nutr. 2010 Mar-Apr;34(2):156-9. doi: 10.1177/0148607110361910. PMID 20375423
- [Result] Pichard C, Kyle UG, Morabia A, Perrier A, Vermeulen B, Unger P. Nutritional assessment: lean body mass depletion at hospital admission is associated with an increased length of stay. Am J Clin Nutr. 2004 Apr;79(4):613-8. doi: 10.1093/ajcn/79.4.613. PMID 15051605
- [Result] Yasunaga H, Horiguchi H, Matsuda S, Fushimi K, Hashimoto H, Ayanian JZ. Body mass index and outcomes following gastrointestinal cancer surgery in Japan. Br J Surg. 2013 Sep;100(10):1335-43. doi: 10.1002/bjs.9221. PMID 23939845
- [Result] Schiesser M, Kirchhoff P, Muller MK, Schafer M, Clavien PA. The correlation of nutrition risk index, nutrition risk score, and bioimpedance analysis with postoperative complications in patients undergoing gastrointestinal surgery. Surgery. 2009 May;145(5):519-26. doi: 10.1016/j.surg.2009.02.001. Epub 2009 Mar 27. PMID 19375611
- [Result] Pablo AM, Izaga MA, Alday LA. Assessment of nutritional status on hospital admission: nutritional scores. Eur J Clin Nutr. 2003 Jul;57(7):824-31. doi: 10.1038/sj.ejcn.1601616. PMID 12821882
- [Result] Buzby GP, Knox LS, Crosby LO, Eisenberg JM, Haakenson CM, McNeal GE, Page CP, Peterson OL, Reinhardt GF, Williford WO. Study protocol: a randomized clinical trial of total parenteral nutrition in malnourished surgical patients. Am J Clin Nutr. 1988 Feb;47(2 Suppl):366-81. doi: 10.1093/ajcn/47.2.366. PMID 3124598
- [Result] Veterans Affairs Total Parenteral Nutrition Cooperative Study Group. Perioperative total parenteral nutrition in surgical patients. N Engl J Med. 1991 Aug 22;325(8):525-32. doi: 10.1056/NEJM199108223250801. PMID 1906987
- [Result] Sungurtekin H, Sungurtekin U, Hanci V, Erdem E. Comparison of two nutrition assessment techniques in hospitalized patients. Nutrition. 2004 May;20(5):428-32. doi: 10.1016/j.nut.2004.01.006. PMID 15105029
- [Result] Oh CA, Kim DH, Oh SJ, Choi MG, Noh JH, Sohn TS, Bae JM, Kim S. Nutritional risk index as a predictor of postoperative wound complications after gastrectomy. World J Gastroenterol. 2012 Feb 21;18(7):673-8. doi: 10.3748/wjg.v18.i7.673. PMID 22363139
- [Result] Keys A, Fidanza F, Karvonen MJ, Kimura N, Taylor HL. Indices of relative weight and obesity. Int J Epidemiol. 2014 Jun;43(3):655-65. doi: 10.1093/ije/dyu058. Epub 2014 Apr 1. PMID 24691951
- [Result] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Result] Kulig J, Sierzega M, Kolodziejczyk P, Dadan J, Drews M, Fraczek M, Jeziorski A, Krawczyk M, Starzynska T, Wallner G; Polish Gastric Cancer Study Group. Implications of overweight in gastric cancer: A multicenter study in a Western patient population. Eur J Surg Oncol. 2010 Oct;36(10):969-76. doi: 10.1016/j.ejso.2010.07.007. Epub 2010 Aug 21. PMID 20727706
- See also: WHO fact sheet — http://www.who.int/news-room/fact-sheets/detail/malnutrition